CLINICAL TRIAL: NCT03864055
Title: Otogenic Cerebral Sinus Vein Thrombosis in Children: Retrospective Case Series and Associated Thrombophilia
Brief Title: Otogenic CSVT Retrospective Case Series and Associated Thrombophilia
Acronym: CSVT PCR
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Kfir Siag, Dr. Siag Kfir, HaEmek Medical Center, Israel
Other Study IDs: 108-18-EMC
Record Dates: First submitted 2019-02-23; First posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Lateral Sinus Thrombosis; Mastoiditis; Otitis Media
Keywords: otitis media; mastoiditis; Lateral Sinus Thrombosis; subperiosteal abscess; sigmoid sinus; mastoid; mastoidectomy; ventilation tube
MeSH Terms: conditions — Lateral Sinus Thrombosis; Mastoiditis; Otitis Media

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — cultures from blood, ear secretions and samples collected during a surgical procedure. also PCR (polymerase chain reaction assay) analysis for bacterial RNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Otogenic CSVT: Children with Otogenic Cerebral Sinus Vein Thrombosis (CSVT)

SUMMARY:
The aim of this study is to report the clinical presentation, Microbiological, laboratory and imaging evaluation, prothrombotic factors analysis, medical and surgical management and outcomes in children with Otogenic Cerebral Sinus Vein Thrombosis (CSVT).

DETAILED DESCRIPTION:
Objective: Otogenic Cerebral Sinus Vein Thrombosis (CSVT) is a rare but serious intracranial complication of otitis media in children. The aim of this study is to report the clinical presentation, Microbiological, laboratory and imaging evaluation, prothrombotic factors analysis, medical and surgical management and outcomes in children with otogenic CSVT. Study design: Retrospective case series

ELIGIBILITY:
Inclusion Criteria:

* age of 18 years or younger
* both sexes are included
* a clinical or radiological finding of mastoiditis in the patient's file
* Documentation of CSVT in an imaging study, either CT or MRI.

Patient's exclusion criteria

* age above 18 years
* lack of a clinical or radiological finding of mastoiditis in the patient's file
* Lack of documentation of CSVT in an imaging study, either CT or MRI.
* previous unprovoked venous thromboembolism event.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with otogenic CSVT
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2018-12-02 (Actual); Primary Completion 2019-02-03 (Actual); Study Completion 2019-02-03 (Actual)

PRIMARY OUTCOMES:
Clinical Presentation | All cases and follow up documentation reported up to a designated date 31 August 2018 predetermined by the institutional ethics committee
  Clinical presentation signs and symptoms will be collected and a summary will be represented in a table including all subjects
Cultures result | All cases and follow up documentation reported up to a designated date 31 August 2018 predetermined by the institutional ethics committee
  the results of cultures from blood, ear secretions, surgery samples, and PCR(polymerize chain reaction assay) will be summarized for the percentage of each pathogen and number of positive results from each type of test
Morbidity and Mortality | All cases and follow up documentation reported up to a designated date 31 August 2018 predetermined by the institutional ethics committee
  The percentage of Morbidity and Mortality until the end of the follow-up period. Morbidity will include any long term sequelae including permanent neurological deficits, chronic ear inflammation, recurrent mastoiditis, and recurrent thromboembolic events.
Surgical intervention | All cases and follow up documentation reported up to a designated date 31 August 2018 predetermined by the institutional ethics committee
  Summary of all surgical interventions, and determination of the common types of surgery performed.
Thrombophilia evaluation tests | All cases and follow up documentation reported up to a designated date 31 August 2018 predetermined by the institutional ethics committee
  Thrombophilia evaluation test results will be collected and a summary will be represented in a table including all subjects

SECONDARY OUTCOMES:
Imaging Studies results | All cases and follow up documentation reported up to a designated date 31 August 2018 predetermined by the institutional ethics committee
  Common diagnosis and distribution of CSVT as mentioned by the radiologist's reports

CONTACTS AND LOCATIONS:
Overall Officials: Kfir Siag, MD, Principal Investigator — haemek medical center
Locations (1):
- HaEmek Medical Center, Afula, Israel

REFERENCES:
- [Background] Ichord R. Cerebral Sinovenous Thrombosis. Front Pediatr. 2017 Jul 27;5:163. doi: 10.3389/fped.2017.00163. eCollection 2017. PMID 28798906
- [Background] Skinner R, Koller K, McIntosh N, McCarthy A, Pizer B; United Kingdom Children's Cancer Study Group (UKCCSG); Paediatric Oncology Nursing Forum (PONF) Supportive Care Group. Prevention and management of central venous catheter occlusion and thrombosis in children with cancer. Pediatr Blood Cancer. 2008 Apr;50(4):826-30. doi: 10.1002/pbc.21332. PMID 17729250
- [Background] Schneider S, Kapelushnik J, Kraus M, El Saied S, Levi I, Kaplan DM. The association between otogenic lateral sinus thrombosis and thrombophilia - A long-term follow-up. Am J Otolaryngol. 2018 May-Jun;39(3):299-302. doi: 10.1016/j.amjoto.2018.03.013. Epub 2018 Mar 7. PMID 29530427
- [Background] Kenet G, Waldman D, Lubetsky A, Kornbrut N, Khalil A, Koren A, Wolach B, Fattal A, Kapelushnik J, Tamary H, Yacobovitch J, Raveh E, Revel-Vilk S, Toren A, Brenner B. Paediatric cerebral sinus vein thrombosis. A multi-center, case-controlled study. Thromb Haemost. 2004 Oct;92(4):713-8. doi: 10.1160/TH04-03-0182. PMID 15467900
- [Background] Zanoletti E, Cazzador D, Faccioli C, Sari M, Bovo R, Martini A. Intracranial venous sinus thrombosis as a complication of otitis media in children: Critical review of diagnosis and management. Int J Pediatr Otorhinolaryngol. 2015 Dec;79(12):2398-403. doi: 10.1016/j.ijporl.2015.10.059. Epub 2015 Nov 5. PMID 26590005
- [Background] Novoa E, Podvinec M, Angst R, Gurtler N. Paediatric otogenic lateral sinus thrombosis: therapeutic management, outcome and thrombophilic evaluation. Int J Pediatr Otorhinolaryngol. 2013 Jun;77(6):996-1001. doi: 10.1016/j.ijporl.2013.03.030. Epub 2013 Apr 29. PMID 23639339
- [Background] Kenet G, Kirkham F, Niederstadt T, Heinecke A, Saunders D, Stoll M, Brenner B, Bidlingmaier C, Heller C, Knofler R, Schobess R, Zieger B, Sebire G, Nowak-Gottl U; European Thromboses Study Group. Risk factors for recurrent venous thromboembolism in the European collaborative paediatric database on cerebral venous thrombosis: a multicentre cohort study. Lancet Neurol. 2007 Jul;6(7):595-603. doi: 10.1016/S1474-4422(07)70131-X. PMID 17560171
- [Background] Kvaerner KJ, Bentdal Y, Karevold G. Acute mastoiditis in Norway: no evidence for an increase. Int J Pediatr Otorhinolaryngol. 2007 Oct;71(10):1579-83. doi: 10.1016/j.ijporl.2007.06.022. Epub 2007 Aug 20. PMID 17707917
- [Background] deVeber G, Andrew M, Adams C, Bjornson B, Booth F, Buckley DJ, Camfield CS, David M, Humphreys P, Langevin P, MacDonald EA, Gillett J, Meaney B, Shevell M, Sinclair DB, Yager J; Canadian Pediatric Ischemic Stroke Study Group. Cerebral sinovenous thrombosis in children. N Engl J Med. 2001 Aug 9;345(6):417-23. doi: 10.1056/NEJM200108093450604. PMID 11496852
- [Background] Pang LH, Barakate MS, Havas TE. Mastoiditis in a paediatric population: a review of 11 years experience in management. Int J Pediatr Otorhinolaryngol. 2009 Nov;73(11):1520-4. doi: 10.1016/j.ijporl.2009.07.003. Epub 2009 Sep 15. PMID 19758711
- [Background] Palma S, Fiumana E, Borgonzoni M, Bovo R, Rosignoli M, Martini A. Acute mastoiditis in children: the "Ferrara" experience. Int J Pediatr Otorhinolaryngol. 2007 Nov;71(11):1663-9. doi: 10.1016/j.ijporl.2007.06.018. Epub 2007 Aug 2. PMID 17681615